CLINICAL TRIAL: NCT04848896
Title: A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and Effectiveness of REAL INTELLIGENCE™ CORI™ in Total Knee Arthroplasty (TKA) Procedure
Brief Title: Study to Evaluate the Safety and Effectiveness of the REAL INTELLIGENCE™ CORI™ in Total Knee Arthroplasty (TKA) Procedure
Acronym: CORI RCT TKA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CORI.2020.08
Record Dates: First submitted 2021-04-07; First posted 2021-04-19 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Arthroplasty; Replacement; Knee
Keywords: Osteoarthritis; Total Knee Arthroplasty (TKA)
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CORI (Experimental): Subjects in need for total knee arthroplasty (TKA) as decided by their doctor and treated with CORI Robotics System.
  Interventions: Device: CORI Robotics
- Conventional Procedure (Active Comparator): Subjects in need for total knee arthroplasty (TKA) as decided by their doctor and treated with conventional approach with conventional manual instrumentation.
  Interventions: Procedure: Conventional Procedure

INTERVENTIONS:
Device: CORI Robotics — Total knee arthroplasty (TKA) treated with CORI Robotics System.
  Arms: CORI
Procedure: Conventional Procedure — Total knee arthroplasty (TKA) treated with conventional approach with conventional manual instrumentation.
  Arms: Conventional Procedure

SUMMARY:
Background:

REAL INTELLIGENCE™ CORI™ (CORI Robotics) is a computer-assisted orthopaedic surgical navigation and burring system. CORI Robotics is designed to help surgeons in planning and executing certain types of knee surgery involving bone preparation. These types of surgery are called 'unicondylar knee arthroplasty' (UKA) and 'total knee arthroplasty' (TKA).

Purpose:

This study is being carried out to demonstrate the safety and effectiveness of the CORI Robotics in TKA procedure. The data collected will be used to demonstrate the safety and effectiveness of CORI and to register CORI in China mainland. The primary objective of this study is to evaluate the use of CORI in TKA procedure in achieving post-operative leg alignment as compared to procedures using conventional manual instruments.

Research participants / locations:

140 research participants will be recruited from up to 8 sites in 3 countries globally (Australia, China Mainland, Hong Kong and New Zealand). There will be 70 patients having TKA using CORI and 70 patients having TKA using conventional procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a suitable candidate for a TKA procedure using CORI and a corresponding S+N Knee Implant System.
2. Subject requires a cemented TKA as a primary indication that meets any of the following condition:

   * Non-inflammatory degenerative joint disease, including osteoarthritis
   * Rheumatoid arthritis
   * Avascular necrosis
   * Requires correction of functional deformity
   * Requires treatment of fractures that were unmanageable using other techniques
3. Subject is of legal age to consent and considered skeletally mature (≥ 18 years of age at the time of surgery)
4. Subject agrees to consent to and to follow the study visit schedule (as defined in the study protocol and informed consent form), by signing the Ethical Committee (EC) or Institutional Review Board (IRB) approved informed consent form.
5. Subject plans to be available through two (2) year postoperative follow-up.
6. Applicable routine radiographic assessment is possible.

Exclusion Criteria:

1. Subject requires a TKA on the index joint as a revision for a previously failed surgery, or has the need for complex implants, or any other implant than a standard TKA (e.g. stems, augments, or custom-made devices).
2. Subject has been diagnosed with post-traumatic arthritis.
3. Subject receives simultaneous bilateral UKA OR a unilateral UKA with contralateral TKA.
4. Subject has one or more of the following arthroplasties that are not fully healed and well-functioning, as determined by the investigator:-Contralateral primary TKA or UKA, however, the subject can only have one knee enrolled in this study.
5. Subject does not understand the language used in the Informed Consent Form.
6. Subject does not meet the indication or is contraindicated for TKA according to the specific Smith+Nephew Knee System's Instructions For Use (IFU).
7. Subject has active infection or sepsis (treated or untreated).
8. Subject is morbidly obese with a body mass index (BMI) greater than 40.
9. Subject is pregnant or breast feeding at the time of surgery.
10. Subject, in the opinion of the Investigator, has advanced osteoarthritis or joint disease at the time of surgery and was better suited for an alternate procedure.
11. Subject currently enrolled in another orthopedic clinical trial study.
12. Subject has a condition(s) that may interfere with the TKA survival or outcome (i.e., Paget's or Charcot's disease, vascular insufficiency, muscular atrophy, uncontrolled diabetes, moderate to severe renal insufficiency or neuromuscular disease, or an active, local infection).
13. Subject in the opinion of the Investigator has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study including mental illness, intellectual disability, drug or alcohol abuse.
14. Subject, in the opinion of the Investigator, has a neuromuscular disorder that prohibited control of the index joint.
15. Subject is a prisoner or meets the definition of a Vulnerable Subject per International Organization for Standardization (ISO) 14155:2020 Section 3.55.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-02-12 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
Post-operative Leg Alignment | 6 weeks
  Post-operative leg alignment via radiographic assessment. Post-operative leg alignment is achieved when the deviation from the subject specific target does not exceed ±3 degrees.

SECONDARY OUTCOMES:
Component Alignment | 6 weeks
  Component alignment will be assessed on long leg standing antero-posterior (A/P) X-rays and standard non weight bearing lateral X-rays taken 6 weeks after surgery
Radiographic Assessment | 12 months and 24 months
  Radiographic assessment on antero-posterior (A/P) and lateral (L) views shall be performed to identify the presence of radiolucent lines, osteolysis & implant migration.
2011 Knee Society Score (KSS) | Pre-op, 6 weeks, 6 months, 12 months and 24 months
  The Functional Knee Score is derived from assessments of walking and standing, standard activities, advanced activities, and discretionary activities in TKA subjects. The 2011 Knee Society Score consists of 4 separate subscales:
  1. An "Objective" Knee Score (seven items: 100 points)
  2. A Patient Satisfaction Score (five items: 40 points)
  3. A Patient Expectation Score (three items: 15 points)
  4. A Functional Activity Score (19 items: 100 points).
  A higher number is a better outcome.
Oxford Knee Score (OKS) | Pre-op, 6 weeks, 6 months, 12 months and 24 months
  To specifically assess the patient's perspective of outcome following knee arthroplasty surgery in TKA subjects. Responses to each question ranges from 0-4 with a range of a possible overall score from 0-48. A score of 0 is the worst possible outcome while a score of 48 is the best possible outcome.
Forgotten Joint Score (FJS) | 6 weeks, 6 months, 12 months and 24 months
  To assess joint-specific patient reported outcomes in TKA subjects. Responses to 12 questions are recorded with a five point Likert response format: "Never", "almost never", "seldom", "sometimes" and "mostly". The item scores are summed and linearly transformed in a 0 to 100 scale and then reversed with a high value reflecting the ability of the subject to forget about the replaced knee joint during the activities of daily living. A score of 100 is the best possible outcome.
EuroQol Five-Dimensional Five-Level (EQ-5D-5L) | Pre-op, 6 weeks, 6 months, 12 months and 24 months
  To assess the subject's health state in TKA subjects. The EQ-5D-5L is composed of the EQ-5D-5L descriptive system and the EQ Visual Analogue scale (EQ VAS). The descriptive system comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Responses are coded as single-digit numbers expressing the severity level selected in each dimension. For instance, 'slight problems' (e.g. 'I have slight problems in walking about') is always coded as '2'. The digits for the five dimensions are combined in a 5-digit code. The EQ- 5D-5L index value is derived by using the vendor supplied calculator to convert each 5-digit EQ-5D-5L profile. The EQ VAS corresponds to a 20 cm vertical, visual analogue scale ranging from 'the best health you can imagine' to 'the worst health you can imagine'. A higher number is a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Lankiewicz, Study Director — Smith & Nephew, Inc.
Locations (4):
- Northern Hospital, Epping, Australia
- Jishuitan Hospital, Beijing, Beijing, China
- The Prince of Wales Hospital, Shatin, Hong Kong
- North Shore Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No